CLINICAL TRIAL: NCT06633653
Title: Mechanism Study of Metabolic Response and Health Benefit Induced by Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE22223R
Record Dates: First submitted 2024-09-25; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- exercise intervention (Experimental)
  Interventions: Behavioral: exercise intervention

INTERVENTIONS:
Behavioral: exercise intervention — Patients will participate in an 8-week supervised aerobic exercise program, the intensity was set at the moderate to vigorous intensity (≥150mins/week exercise on the treadmill).

SUMMARY:
This study is a single-arm, self-control, single-center study to investigate the mechanism under exercise inducing metabolic response and health benefit. 40 overweight/obese patients with prediabetes will be recruited in this study and instructed to participate in an 8-week exercise program. We aim to investigate 1) the changes of phenotypes such as body weight, body fat, laboratory values, appetite, resting energy expenditure, myokine-adipokine before and after exercise 2) the changes of serum metabolomics 3) search for potential biomarkers of exercise through multi-omics integrated analysis of metabolomics, metagenomics, phenomics, single-cell transcriptome, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Han Chinese
2. 5.6 mmol/L≤fasting blood glucose<7 mmol/L, and/or 7.8 mmol/L≤2h-postload glucose<11.1mmol/L, and/or 5.7% ≤HbA1c<6.5% without anti-hyperglycemic medicine treatment
3. Voluntary participation and provide informed consent

Exclusion Criteria:

1. Participated in any clinical study in relation to weight-loss in the past 1 year
2. Had a weight change of more than 10% present weight in the past 1 year
3. Had a drug usage not suitable for this study in the past 3 months, such as hormone drug, orlistat, metformin, GLP-1 receptor agonists, lipid-lowering agents, liver protection drug, etc
4. Presence of diseases influencing glucose and lipid metabolism ,such as hyperthyroidism, hypothyroidism, Cushing syndrome, etc
5. Poorly controlled blood pressure: systolic blood pressure≥180mmHg, and/or diastolic blood pressure≥100mmHg
6. Presence of serious heart, liver, kidney or systemic diseases
7. Presence of skeletal and muscular diseases which make it difficult to exercise
8. Received any kind of surgery in the past 1 year
9. COVID-19 positive or recovery from COVID-19 within 4 weeks
10. Presence of eating disorders or have a history of eating disorders
11. Presence of sleep disorders
12. Work in disrupted circadian rhythms
13. Pregnancy and breastfeeding women

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-09 (Estimated); Primary Completion 2027-10-09 (Estimated); Study Completion 2027-10-09 (Estimated)

PRIMARY OUTCOMES:
Changes of serum metabolites detected by metabolomic profiling | From enrollment to the end of exercise intervention at 8 weeks

SECONDARY OUTCOMES:
Changes of anthropometrics including body weight, body fat, waist-to-hip ratio | From enrollment to the end of exercise intervention at 8 weeks
Changes of laboratory values including plasma glucose, insulin, lipids, liver enzymes, thyroid hormones, inflammation cytokines | From enrollment to the end of exercise intervention at 8 weeks

OTHER OUTCOMES:
Changes of resting energy expenditure | From enrollment to the end of exercise intervention at 8 weeks
Changes of fecal microbial composition detected by metagenomics | From enrollment to the end of exercise intervention at 8 weeks
Changes of serum proteins detected by proteomics | From enrollment to the end of exercise intervention at 8 weeks
Changes of peripheral blood CD45+ cells detected by single cell sequencing | From enrollment to the end of exercise intervention at 8 weeks